CLINICAL TRIAL: NCT06237400
Title: A Phase I/II Dose Escalation and Expansion Study to Evaluating the Tolerability, Safety, Efficacy, and Pharmacokinetics of ZG19018 in Patients With KRAS G12C Mutant Advanced Solid Tumors.
Brief Title: A Study of ZG19018 in Patients With KRAS G12C Mutant Advanced Solid Tumors.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG19018-001
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: KRAS G12C Mutant Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): Dose escalation will begin with rapid dose escalation for the low-dose groups (50 mg QD 、150 mg QD) and a "3 + 3" dose-escalation protocol for the high-dose groups.
  Interventions: Drug: ZG19018
- Phase 2 Dose Expansion (Experimental): Upon completing the dose escalation part of the study, dose expansion may proceed with 3 groups consisting of subjects with KRAS G12C mutant advanced solid tumors，Including non-small cell lung cancer, colorectal cancer and Other advanced solid tumors
  Interventions: Drug: ZG19018

INTERVENTIONS:
Drug: ZG19018 — ZG19018 Given by PO (mouth)

SUMMARY:
Evaluate the safety and tolerability of ZG19018 in Patients with KRAS G12C mutant advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who fully understood this trial and voluntarily signed the informed consent form;
* Men or women ≥ 18 years old;
* ECOG Performance Status (PS) 0 or 1;
* Life expectancy > 3 months.

Exclusion Criteria:

* Received any treatment with inhibitors against KRAS G12C mutation at any time, e.g., AMG 510, MRTX 849, etc.;
* Patients requiring medications that can potentially prolong QTc interval;
* Other conditions that the investigator considers to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 21Days
  A DLT is defined as any Grade ≥ 3 AE meeting the criteria listed below occurring during the first treatment cycle of ZG19018 (day 1 through day 21) where elationship to ZG19018 cannot be ruled out.
Objective Response Rate (ORR) | Up to 24 Months
  The sum of the proportions of subjects who achieved CR or PR in imaging evaluation as assessed by the investigator based on RECIST1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No